CLINICAL TRIAL: NCT02269384
Title: The Effects of Pain and the Memory of Pain on Autonomic and Neuromuscular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mount St. Mary's College, Los Angeles, CA (Other)
Responsible Party: Principal Investigator, Derrick Sueki, Principal Investigator, Mount St. Mary's College, Los Angeles, CA
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MountSMCLA
Record Dates: First submitted 2014-10-11; First posted 2014-10-21 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Pain
Keywords: Pain; Memory; Pressure Pain Threshold; Electromyography; Heart Rate Variability
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- No History of Significant Injury (Sham Comparator): Experimental Noxious Stimulus, Memory of Experimental Noxious Stimulus, Memory of Prior Significant Injury, Mental Challenge Test
  Interventions: Procedure: Experimental Noxious Stimulus; Behavioral: Memory of Experimental Noxious Stimulus; Behavioral: Memory of Prior Significant Injury; Procedure: Mental Challenge Test
- History of Significant Injury (Active Comparator): Experimental Noxious Stimulus, Memory of Experimental Noxious Stimulus, Memory of Prior Significant Injury, Mental Challenge Test
  Interventions: Procedure: Experimental Noxious Stimulus; Behavioral: Memory of Experimental Noxious Stimulus; Behavioral: Memory of Prior Significant Injury; Procedure: Mental Challenge Test

INTERVENTIONS:
Procedure: Experimental Noxious Stimulus — Localized manual pressure will be placed up predetermined points on the lower extremity until maximum pain tolerance levels are reached.
  Other Names: Acute Pain Stimulus
Behavioral: Memory of Experimental Noxious Stimulus — Subjects will be asked to visualize previously experience experimental noxious stimulus
Behavioral: Memory of Prior Significant Injury — Subjects will visual prior significant injury or a predetermined lower extremity region in control subjects.
Procedure: Mental Challenge Test — Subjects will count backwards from 100 by specified amounts as rapidly as possible

SUMMARY:
The prevalence of chronic pain has been estimated at 30% in the US and these values may under report the true prevalence of people who experience long term pain as additional research has shown that 73% will have a reoccurrence of symptoms within 12 months of the original injury indicating that while the pain and symptoms may resolve, additional impairments or issues may underlie the symptoms.

Biopsychosocial factors such as depression, post traumatic stress, anxiety, pain catastrophizing, and negative emotions have been closely linked to pain and can influence a patient's pain perceptions. Along these lines, the memory of past experiences and trauma potentially play a large role in these biopsychosocial responses. Research is evolving and a strong correlation has been established between chronic pain and prior history of trauma or abuse and also non-traumatic incidents such as motor vehicle accidents and injuries/surgical procedures. This has led to speculation and research that explores how a variety of life events may become stimulants for long-term alterations in the processing and manifestation of pain and how they may have an enduring impact on physical health outcomes.

The proposed research will add to the body of knowledge underlying the association between pain, memory, autonomic system, and neuromuscular function. The goal of this project is to study the relationship between pain memory systems, specifically acute pain, short-term memory of pain, and long term pain memory, and their effects upon neuromuscular and autonomic system responses in the body.

DETAILED DESCRIPTION:
Study Design This study will utilize a repeated measures quasi-experimental case control design structure. Subjects will be placed into two groupings, those who have a history of prior lower extremity injury and those who have no history of lower extremity injury. The two groupings will be age and gender matched. Subjects who have no prior history of lower extremity injury will be matched to subjects with a prior history of injury. There will be an equivalent number of participants per group with similar demographic information in both groups in order to reduce the number of variables influencing the results of the experiment. Within each of these groupings, specific interventions will be clustered and performed as a set. These clusters of interventions will be randomized to minimize internal testing error. Both groups of participants will be exposed to the same interventions (baseline, pain pressure, visualization of pain pressure and prior injury, and mental challenge test). Investigators responsible for testing and outcome measurement will be blinded to the groupings of subjects (past history or no prior history of injury). It is anticipated that the testing, including initial set up, will take between 60 and 75 minutes. All testing will take place at the Mount St. Mary's College physical therapy exercise and research lab or in a private room at Knight Physical Therapy Inc.

Study Methods Initial Set Up (25 minutes) Upon commencement of the study, subjects will be asked to fill out the Tampa Kinesiophobia Questionnaire, Fear Avoidance Belief Questionnaire, Fear of Pain Scale, Pain Catastrophizing Scale, and the Vividness of Visual Imagery Questionnaire. This should take approximately 10 minutes. Following completion of these questionnaires, they will be introduced to the investigators and then asked to lie supine upon the treatment table. A pillow will be placed under their head for comfort. Surface EMG rRecording electrodes will be placed upon the belly of the tibialis anterior muscle. An electrode will be placed upon the medial tibia and will serve as a ground for the other two electrodes. Placement of electrodes will correspond to the side of injury (i.e. prior injury to the right ankle would result in electrode placement on the right tibialis anterior and right anterior deltoid muscles). In subjects without history of injury, side of electrode placement will be predetermined and randomized. Also at this time, subjects with a prior history of injury will be asked to identify the location of the injury. The tester will then palpate the area of previous injury and will locate the tender point in this area. This point will be marked with a pen for later use. In subjects with no prior injury, the anterior talofibular ligament, the lateral knee joint line, or the lateral belly of the gastrocnemius muscle will be located and marked on the side of testing. The site will be randomized so as to blind testers. Testers will be informed of the side to be tested through the sealed envelope that is opened prior to testing. They will be blinded as to prior injury grouping.

At this point, the subject will be walked through the procedure and an initial pain pressure threshold measurement will be taken and a simulated break test (see below for description of break test) will be performed at the foot / ankle in order to familiarize the subject with the test procedures and also to ensure that all equipment is functioning optimally. This process should take approximately 10 minutes.

Following this procedure, a timer will be set and the subject will rest in this position for five minutes to acclimate to the environment and to normalize their autonomic system.

Autonomic System Response (10 minutes) Following the five-minute acclimation period, heart rate variability (HRV) data will be recorded, marked, and used as a baseline measurement. The HRV data will be collected throughout each testing procedure. Initially, at the site of previous injury (or randomized pressure site for subjects with no prior history of injury), the tester will use their thumb to apply pressure to the site. The pressure will increase until the subject reports their maximal pain level. Prior to the application of pressure, the subject will be informed that they are to experience the maximum pain tolerable and to inform the tester when that level is reached. The subject will next be instructed to notify the testers when they have reached the maximum tolerable pain. Once achieve, the pressure will be maintained for 10 seconds in order to get a baseline HRV recording. After 10 seconds, the pressure will be released and the HRV recording will be marked. At this time, the subject will be asked to report their level of pain on a scale of 1 to 10. The subject will then rest for three minutes to return their HRV to baseline values. At this point, the subject will be instructed to close their eyes and imagine the pain pressure in their leg that was just applied. HRV and pain values will be marked and recorded. The subject will rest for another three minutes and then they will once again be asked to close their eyes. In this instance, they will be asked to visualize the details of their prior injury. In subjects with no prior injury, they will asked to visualize the muscles, bone, and blood flow of their tibia. Like before, HRV and pain values will be marked and recorded. Following another three minute rest period, the subject will be asked to complete a mental challenge test. This test will require subjects to count backwards as quickly as possible from 100 by 7. HRV and pain values will be marked and recorded. With this test, and with all testing, the subject will be allowed to withdrawal from the test for any reason and without repercussions.

Pressure Pain Threshold (10 minutes) The amount of pain and the force required to elicit the pain response will be applied and monitored by a Wagner Force Ten™ FDX Digital Force Gauge Pain Algometer. The algometer is a device designed to measure sensitiveness to pressure and in pain studies; the algometer is used to measure sensitiveness to pain as a product of pressure. The Wagner Force Ten Digital Algometer is a portable unit with a small 1 cm2-rubberized tip capable of applying pressures up to 50 lbs./ft. The unit is capable of remembering multiple data points and storing peak force and force-averaged data that will be retrieved after testing for later analysis. During each of the five test components (Baseline, Pain Pressure, Visualization of Pain Pressure, Visualization of Prior Injury, and Mental Challenge Test) the testing procedures will be identical to those applied earlier, except instead of measuring muscle performance or HRV, pain pressure will be recorded. The tip of the pain algometer will be placed upon the site of prior injury or upon the anterior talofibular ligament. Pressure will be applied through the algometer and the subject will be instructed to inform the tester when they first begin to experience pain. This value will be recorded along with HRV values.

Neuromuscular Response (15 minutes) During the next phase of testing, a small rolled up towel will be placed under the test ankle. The towel will be utilized to raise the foot from the table in order to facilitate testing. At this point, the tester will stabilize the lower extremity by grasping the calf approximately 12 inches above the malleolus. This hand will provide a counter force to the forces applied by the test hand. In the test hand, a Hoggan Scientific Microfet 2TM Handheld Muscle Tester will be placed upon the lateral aspect of the fifth metatarsal bone of the foot. The placement will be proximal on the metatarsal approximately at the base of the fifth metatarsal bone. The position of the sensor will be marked to standardize test position and measured for later force measurement purposes. The subject will be instructed to isometrically resist the force applied by the tester. At this point, Surface EMG and Force recording will commence simultaneously. The Surface EMG will be utilized to measure action potential propagation. Surface recording electrodes are placed upon the skin to measure these action potentials. At no time will needles be utilized to collect data and therefore, no penetration of the skin is required. The initiation of the test will also be noted on the HRV recording. A steady but increasing amount of force will be applied slowly and gradually to the foot in a medially and slightly caudal direction until the subject can no longer resist the force. This process is called the "break test" because the muscle is tested until it can no longer resist the force. The subject will rest for 30 seconds after which the break test and associated data recordings will be repeated two more times with a 30-second rest period in between tests.

The subject will be allowed to rest for three minutes prior to beginning the next portion of the study. HRV testing will be started and then the tester as previously described will place pain pressure upon the site of previous injury. The location of this site has been previous marked for consistency of application. In subjects with no prior history of injury, the pressure will be applied to the anterior talofibular ligament. When pain pressure has reached it's maximal levels, a second tester will perform a break test on the subject. Following the test, the subject will rest for 30 seconds and the process will be repeated two more times with a 30 second rest period in between tests. Force, EMG, HRV, and pain values will be recorded during each of the break tests.

Following a three minute rest period, the subject will asked to visualize the pain pressure placed upon the leg (or visualize their tibia as previously described) and three break tests will be performed during the visualization process. Force, EMG, HRV, and pain values will be recorded during each of the break tests. This process will be repeated for visualization of prior injury and for the mental challenge test.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have experienced a significant injury in the lower extremity (i.e. fracture, ligament strain, surgery, trauma) that resulted in a significant loss of function for greater then three weeks time period will be included in the study.
* Significant loss of function will be defined as not being able to walk or being required to use crutches for the three weeks and trauma shall be defined as physical, emotional, or social distress or suffering that also coincided with injury to the lower extremity.
* Individuals with a history of significant injury to the lower extremity will be age and gender matched with individuals who have no history of traumatic injury.

Exclusion Criteria:

* Acute injuries in the lower extremity occurring less than six weeks prior,
* any heart conditions, any open wounds in their lower extremities,
* severe hypertension greater than 180/110,
* poor sensation in the lower extremities, or
* cognitive impairments that prevent following the instructions of the study, and
* chronic pain greater then 3/10 in any region of the body.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Change in surface electromyography (sEMG) from baseline to either during or immediately post intervention or condition | Data will be collected in one, one hour session. During the session, sEMG will be collected during or immediately following intervention or condition.
  Surface electrodes will be placed upon the tibialis anterior muscle to monitor muscle activity during testing.
Change in hand held dynamometric (HHD) measures from baseline to either during or immediately post intervention or condition | Data will be collected in one, one hour session. During the session, HHD will be collected during or immediately following intervention or condition
  A Hoggan Scientific Microfet 2 Handheld Muscle Tester will be placed upon the lateral aspect of the fifth metatarsal bone of the foot and a plantar and eversion directed force will be applied until the muscle can no longer resist the force applied (break test).
Change in pressure pain threshold (PPT) from baseline to either during or immediately post intervention or condition | Data will be collected in one, one hour session. During the session, PPT will be collected during or immediately following intervention or condition
  The force required to elicit the pain response will be applied and monitored by a Wagner Force Ten™ FDX Digital Force Gauge Pain Algometer.
Change in heart rate variability (HRV) from baseline to either during or immediately post intervention or condition | Data will be collected in one, one hour session. Continuous monitoring of HRV will occur during each intervention or condition and significant data points will be marked for future analysis.
  The HRV Live heart rate variability monitoring systems will be utilized and recording sensors will be placed upon the wrist of both arms to monitor cardiovagal responses during testing.

SECONDARY OUTCOMES:
Change in verbal numeric pain scale (NPS) rating from baseline to immediately post intervention or condition | Data will be collected in one, one hour session. During the session, NPS will be collected immediately following intervention or condition.
  Verbal numeric pain scale will be used to monitor the amount of pain the subject is experiencing at various points throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: M. Samuel Cheng, DSc, Study Chair — Nova Southeastern University
Locations (1):
- Mount St. Mary's College, Los Angeles, California, United States

REFERENCES:
- [Derived] Sueki DG, Dunleavy K, Puentedura EJ, Heard L, Van der Heide P, Cheng MS. Differing Effects of Nociception and Pain Memory on Isometric Muscle Strength in Participants With and Without a History of Injury: A Quasi-Experimental Study. Am J Phys Med Rehabil. 2023 Sep 1;102(9):787-794. doi: 10.1097/PHM.0000000000002205. Epub 2023 Feb 3. PMID 36753453